CLINICAL TRIAL: NCT06397482
Title: A Single-Arm, Pilot Study to Assess the Effects of an Encapsulated Calcium Butyrate Dietary Supplement on Gut Health
Brief Title: Effects of an Encapsulated Calcium Butyrate Dietary Supplement on Gut Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kemin Foods LC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BIO-2314
Record Dates: First submitted 2024-04-17; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Healthy; Gastrointestinal Discomfort
Keywords: Butyrate; Butyric Acid; Short-Chain Fatty Acid; Permeability

STUDY DESIGN:
Intervention Model Description: Single-Arm, Pilot Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Encapsulated Calcium Butyrate (Experimental): Subjects will be instructed to consume one 600 mg capsule daily, on an empty stomach, at least 30 minutes before their first meal.
  Interventions: Dietary Supplement: Encapsulated Calcium Butyrate

INTERVENTIONS:
Dietary Supplement: Encapsulated Calcium Butyrate — Contains at minimum 35% butyric acid

SUMMARY:
The primary objective of this single-arm pilot study is to investigate the effects of an encapsulated calcium butyrate dietary supplement on gastrointestinal (GI) health outcomes in healthy adults, including GI symptom severity (e.g., gas/flatulence and abdominal bloating), bowel habits (frequency and consistency), digestion-associated quality of life, and measures of GI permeability.

DETAILED DESCRIPTION:
This will be a single-arm pilot study consisting of one screening visit (day -8) and four intervention visits (days 0, 1, 43, and 44).

On visit 1 (day -8), subjects will arrive at the clinic in a fasting state. After providing voluntary informed consent, subjects will undergo a medical history evaluation along with clinic visit procedures. Blood samples will be collected for safety analyses. Subjects will complete the Gastrointestinal Symptom Rating Scale (GSRS) and the Diet ID questionnaire. A Bowel Habits Diary (BHD) and stool collection kit will be dispensed to complete prior to visit 2.

On visit 2 (day 0), subjects will arrive at the clinic in a fasting state and undergo clinic visit procedures. Fecal samples and the BHD from visit 1 will be collected. Subjects will be administered the GSRS for determination of eligibility (at least mild symptoms of indigestion at visit 1 and 2). Enrolled participants will be administered the Digestion-associated Quality of Life Questionnaire (DQLQ). Blood samples will be collected for markers of intestinal permeability. Subjects will then complete an intestinal permeability test where they will ingest two sugar probes and be instructed to collect all urine over the following 24 h. A BHD and stool collection kit will be dispensed to complete prior to visit 4. Study product and a study product log will be dispensed.

On visit 3 (day 1), subjects will arrive at the clinic to return their urine collection containers.

On visit 4 (day 43), subjects will arrive at the clinic in a fasting state and undergo clinic visit procedures. Fecal samples and the BHD from visit 2 will be collected. Subjects will be administered the GSRS and DQLQ. Blood samples will be collected for safety analyses and markers of intestinal permeability. Subjects will then complete an intestinal permeability test as previously described. The study product log and unused study product will be collected.

On visit 5 (day 44), subjects will arrive at the clinic to return their urine collection containers.

Subjects will receive an email link for an electronic GSRS and DQLQ to be completed on days 8, 15, 22, 29, and 36.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 to ≤60 years of age at visit 1.
2. BMI ≥18.0 and <32.0 kg/m2 at visit 1.
3. A mean ≥3 (at least mild symptoms) in the indigestion domain from the Gastrointestinal Symptom Rating Scale (GSRS) at both visits 1 (day -8) and 2 (day 0).
4. Habitually consumes a standard American diet as defined by a Diet ID diet quality score of ≤6 (~60 on the Healthy Eating Index [HEI]-2015).
5. Willing to abstain from alcohol consumption and vigorous exercise for 24 hours prior to and following visits 2 (day 0) and 4 (day 43).
6. Non-user or former user (daily use; cessation ≥12 months) of tobacco or nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) within 12 months of visit 1, and has no plans to begin use during the study period.
7. Non-user or former user (daily use; cessation ≥12 months) of any marijuana or hemp products within 12 months of visit 1 and has no plans to use marijuana or hemp products during the study period.
8. Willing to maintain habitual physical activity level throughout the duration of the study with the exception of the 24 h before and after visits 2 and 4 (days 0 and 43).
9. Willing to maintain habitual dietary patterns throughout the duration of the study, including stable intake of current vitamins, minerals, supplements, and medications not interfering with study outcomes.
10. Female subject who is willing to wear a tampon during the stool and urine collection if the collection occurs during menstruation.
11. No health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator based on medical history.
12. Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Known sensitivity, intolerability, or allergy to any of the study products or their excipients.
2. Abnormal laboratory test results of clinical significance at visit 1 (day -8), at the discretion of the Clinical Investigator. One re-test will be allowed on a separate day prior to visit 2 (day 0), for subjects with abnormal laboratory test results.
3. Clinically important GI condition that would potentially interfere with the evaluation of the study product (e.g., inflammatory bowel disease, irritable bowel syndrome, Crohn's disease, celiac disease, history of surgery for weight loss, gastroparesis, and clinically significant lactose or gluten intolerance or other food or ingredient allergies).
4. Pre-menopausal female subjects with an irregular menstrual cycle (regular cycle defined as 21 to 35 days in length for the last 3 months prior to visit 1).
5. Recent (within 2 weeks of visit 1; day -8) history of an episode of acute GI illness such as nausea/vomiting or diarrhea (defined as ≥3 loose or liquid stools/d).
6. Self-reported history (within 6 weeks of visit 1; day -8) of constipation (defined as fewer than three bowel movements per week).
7. Uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), hepatic, renal, endocrine (including Type 1 and Type 2 diabetes mellitus), hematologic, immunologic, neurologic (such as Alzheimer's or Parkinson's disease), psychiatric (including depression and/or anxiety disorders) or biliary disorders. Conditions that are well-controlled or resolved will be assessed by the Clinical Investigator on a case-by-case basis.
8. Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at visit 1 (day -8; section 6.3.1).
9. Unstable use (initiation or change in dose) within 1 month of visit 1 (day -8) of FDA-approved medications for hypertension.
10. History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
11. Major trauma or any other surgical event within 3 months of visit 1 (day -8).
12. Signs or symptoms of an active infection of clinical relevance within 5 days of visit 1 (day -8). The visit may be rescheduled once all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to visit 1 (day -8).
13. Weight loss or gain >4.5 kg in the 3 months prior to visit 1 (day -8).
14. Currently or planning to be on a weight loss regimen during the study.
15. Antibiotic use within 1 month of visit 1 (day -8) and throughout the study period.
16. Use of steroids within 1 month of visit 1 (day -8) and throughout the study period.
17. Regular use (i.e., >3 days/week) of anti-inflammatory medications (e.g., NSAIDs) within 1 month of visit 1 (day -8).
18. Use of medications (over-the-counter or prescription) and/or dietary supplements, known to influence GI function, including but not limited to, pre-, post-, and probiotic supplements, fiber supplements, laxatives, enemas, suppositories, H2 blockers, proton pump inhibitors, antacids, anti-diarrheal agents, anti-depressants, and/or anti-spasmodic within 2 weeks of visit 1 (day -8) and throughout the study period. Standard multivitamin and mineral supplements are allowed.
19. Underwent an endoscopy or colonoscopy preparation within 3 months prior to visit 1 (day -8).
20. Exposure to any non-registered drug product within 1 month prior to visit 1 (day -8).
21. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. Subjects who are pregnant during the study will be discontinued.
22. Recent history (within 12 months visit 1; day -8) of alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
23. Self-report of blood donation totaling between 101 mL to 449 mL of blood within 1 month prior to screening or a blood donation of more than 450 mL within 56 days prior to baseline.
24. Receipt or use of study products in another research study within 28 days prior to visit 2 (day 0) or longer if the previous study product is deemed by the Clinical Investigator to have lasting effects that might influence the eligibility criteria or outcomes of the current study.
25. Has a condition the Clinical Investigator believes would interfere with his ability to provide informed consent, and comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Indigestion Symptom Severity | Change from baseline (day 0) to end of each week (day 8, 15, 22, 29, 36, and 43)
  Assessed by the Gastrointestinal Symptom Rating Scale (GSRS): minimum = 1 (no discomfort); maximum = 7 (very severe discomfort)

SECONDARY OUTCOMES:
Other Gastrointestinal Symptom Severity | Change from baseline (day 0) to end of each week (day 8, 15, 22, 29, 36, and 43)
  Abdominal pain, reflux, diarrhea, and constipation assessed by the Gastrointestinal Symptom Rating Scale (GSRS): minimum = 1 (no discomfort); maximum = 7 (very severe discomfort)
Digestion-associated Quality of Life | Change from baseline (day 0) to end of each week (day 8, 15, 22, 29, 36, and 43)
  Assessed by the Digestion-associated Quality of Life Questionnaire (DQLQ): minimum = 0% (never); maximum = 100% (always)
Ease of Stool Passage | Change from baseline (day 0) to end of intervention (day 43)
  Assessed by the Bowel Habits Diary (BHD): minimum = 1 (very easy); maximum = 5 (very difficult)
Stool Consistency | Change from baseline (day 0) to end of intervention (day 43)
  Assessed by the Bristol Stool Scale (BSS): minimum = 1 (very solid); maximum = 7 (entirely liquid)
Intestinal Permeability Marker 1 | Change from baseline (day 0) to end of intervention (day 43)
  Assessed by lactulose/13C mannitol excretion
Intestinal Permeability Marker 2 | Change from baseline (day 0) to end of intervention (day 43)
  Assessed by blood lipopolysaccharide binding protein (LBP) concentrations
Intestinal Permeability Marker 3 | Change from baseline (day 0) to end of intervention (day 43)
  Assessed by blood zonulin concentrations
Fecal Microbiome | Change from baseline (day 0) to end of intervention (day 43)
  Assessed by shotgun metagenomic sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Shah, MD, Principal Investigator — Biofortis Innovation Services
Locations (1):
- Biofortis Innovation Services, Addison, Illinois, United States